CLINICAL TRIAL: NCT02071251
Title: A Study to Evaluate a Quality Improvement Intervention to Reduce Wound Separation Rates in Obese Gynecologic Oncology Service Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108303
Record Dates: First submitted 2014-02-22; First posted 2014-02-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Wound Complications; Wound Infection; Wound Separation
Keywords: Wound complications; Wound infection; Wound separation
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective intervention (Experimental): The skin and subcutaneous tissues were incised using a scalpel or cutting electrocautery. Use of coagulation current on the skin or subcutaneous tissues was not allowed, except focally to attain hemostasis. At the conclusion of surgery, a 7mm Jackson-Pratt drain was placed below Camper's fascia, which in turn was closed with 3-0 plain catgut suture. The skin was closed with staples. Dressings were retained for at least twenty-four hours. Staples were to be retained for at least two weeks.
  Interventions: Procedure: Prospective wound complication protocol

INTERVENTIONS:
Procedure: Prospective wound complication protocol — The skin and subcutaneous tissues were incised using a scalpel or cutting electrocautery. Use of coagulation current on the skin or subcutaneous tissues was not allowed, except focally to attain hemostasis. At the conclusion of surgery, a 7mm Jackson-Pratt drain was placed below Camper's fascia, which in turn was closed with 3-0 plain catgut suture. The skin was closed with staples. Dressings were retained for at least twenty-four hours. Staples were to be retained for at least two weeks.

SUMMARY:
Approximately 500,000 surgical site infections occur annually in the US. These lead to worse patient quality of life, more outpatient and emergency room visits, readmissions and home services, with an estimated increase in costs of at least $3500 per complication. Surgical site infections are associated with increasing body mass index. There is limited and conflicting data of the utility of multiple surgical interventions to decrease the risk of surgical site complications. The investigators explored the effect of a prospective care pathway for closure of vertical abdominal wounds on patient's wound complications.

ELIGIBILITY:
Inclusion Criteria:

Women were eligible if they were between the ages of 18-89, with a BMI ≥ 30 kg/m2 undergoing a gynecologic procedure via a vertical abdominal incision. -

Exclusion Criteria:

Planned laparoscopic surgery, planned panniculectomy or other plastic surgery procedure at the time of laparotomy, prior history of hernia repair with mesh or planned mesh hernia repair at the current procedure, enterotomy or intestinal surgery, a history of prior radiation to the abdomen or pelvis, concurrent pregnancy, current incarceration, or inability to provide informed consent, including inability to understand spoken English.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Wound complication | Within 8 weeks of surgery
  The primary outcome for our study was a wound complication within eight weeks of laparotomy. Wound complication was defined as seroma, hematoma, separation, or infection requiring additional medical and/or surgical management within eight weeks of laparotomy.

SECONDARY OUTCOMES:
Wound separation | 8 weeks of surgery
  Wound separation within 8 weeks of surgery
Wound infection | 8 weeks of surgery
  Wound infection within 8 weeks of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Akiva P Novetsky, MD, MS, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine and Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Bratzler DW, Houck PM; Surgical Infection Prevention Guideline Writers Workgroup. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Am J Surg. 2005 Apr;189(4):395-404. doi: 10.1016/j.amjsurg.2005.01.015. PMID 15820449
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046